CLINICAL TRIAL: NCT01593046
Title: A Randomized, Open Label Study to Investigate the Safety, Tolerability and Pharmacokinetics of Repeat Dose Administration of Long-Acting GSK1265744 and Long-Acting TMC278 Intramuscular and Subcutaneous Injections in Healthy Adult Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Repeat Dose Administration of Long-Acting GSK1265744 and Long-Acting TMC278 Intramuscular and Subcutaneous Injections in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 115428
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK1265744 LAP; integrase inhibitor; healthy subjects; TMC278 LA; GSK1265744LAP; long acting retroviral; HIV-1 infection
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — cabotegravir; Injections, Intramuscular; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Run-in Period (Experimental): Oral GSK1265744 30mg once daily for 14 days
  Interventions: Drug: GSK1265744 Oral
- Cohort 1 (Experimental): GSK1265744 LAP injection given subcutaneously once a month for 4 months
  Interventions: Drug: GSK1265744 LAP 800mg intramuscular injection; Drug: GSK1265744 LAP 200mg subcutaneous injection
- Cohort 2 (Experimental): GSK1265744 LAP injection given intramuscularly once a month for 4 months. TMC278 LA + GSK1265744 given in Month 3 and 4.
  Interventions: Drug: GSK1265744 LAP 800mg intramuscular injection; Drug: GSK1265744 LAP 200mg intramuscular injection; Drug: TMC278 LA 1200mg intramuscular injection; Drug: TMC278 LA 600mg intramuscular injection
- Cohort 3 (Experimental): GSK1265744 LAP injection given intramuscularly once a month for 4 months. TMC278 LA + GSK1265744 given in Month 3 and 4.
  Interventions: Drug: GSK1265744 LAP 800mg intramuscular injection; Drug: GSK1265744 LAP 400mg intramuscular injection; Drug: TMC278 LA 1200mg intramuscular injection; Drug: TMC278 LA 600mg intramuscular injection
- Cohort 4 (Experimental): GSK1265744 LAP injection given intramuscularly once every 12 weeks.
  Interventions: Drug: GSK1265744 LAP 800mg intramuscular injection

INTERVENTIONS:
Drug: GSK1265744 Oral — 30mg tablet
  Other Names: GSK1265744
  Arms: Run-in Period
Drug: GSK1265744 LAP 800mg intramuscular injection — 800mg Loading dose given at month 1 dose
  Other Names: GSK1265744
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: GSK1265744 LAP 200mg subcutaneous injection — 200mg maintenance dose give at months 2 - 4
  Other Names: GSK1265744
  Arms: Cohort 1
Drug: GSK1265744 LAP 200mg intramuscular injection — 200mg maintenance dose given at months 2 - 4
  Other Names: GSK1265744
  Arms: Cohort 2
Drug: GSK1265744 LAP 400mg intramuscular injection — 400mg maintenance dose given at month 2 - 4
  Other Names: GSK1265744
  Arms: Cohort 3
Drug: TMC278 LA 1200mg intramuscular injection — 1200mg Loading dose given at month 3
  Other Names: TMC278 LA
  Arms: Cohort 2; Cohort 3
Drug: TMC278 LA 600mg intramuscular injection — 600mg Loading dose given at month 4
  Other Names: TMC278 LA
  Arms: Cohort 2; Cohort 3
Drug: GSK1265744 LAP 800mg intramuscular injection — 800mg dose given quarterly (once every) 12 weeks
  Other Names: GSK1265744
  Arms: Cohort 4

SUMMARY:
LAI115428 is a Phase I, randomized, repeat dose escalation study to determine the safety, tolerability, and PK profile of intramuscular and subcutaneous injections of GSK1265744 in a long acting parenteral (LAP) formulation in healthy subjects. Subjects will be randomized to 3 monthly dosing cohorts and 1 quarterly dosing cohort with either intramuscular or subcutaneous dosing. In the monthly dosing cohorts subjects will receive GSK1265744 alone for 2 months and then in combination with TMC278 long acting parenteral (LA) for 2 months. For the quarterly dosing cohort, 2 quarterly intramuscular doses of GSK1265744 LAP will be given alone. Three dose levels of GSK1265744 will be evaluated partly in combination with TMC278 LA to adequately characterize the GSK1265744 LAP and TMC278 LA safety, tolerability, and PK profile. A total enrolment of approximately 40 healthy subjects is planned for this study.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinically significant abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 64 years of age inclusive, at the time of signing the informed consent.
* Females of childbearing potential with a negative pregnancy test (serum or urine) at screen and at Day -21, and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception for six months after the final dose of study drug.
* Body weight greater than or equal to 50 kg for men and greater than or equal to 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* All Study subjects should be counseled on the practice of safer sexual practices including the use of effective barrier methods (e.g. male condom/spermicide).

Exclusion Criteria:

* History of bleeding or clotting disorders including disseminated intravascular coagulation, hemophilia Henoch-Schönlein purpura (allergic purpura), hereditary hemorrhagic telangiectasia, thrombocytopenia, thrombophilia or Von Willebrand's disease.
* High-risk behavior for HIV infection including one of the following risk factors within six months before entering the study (day 1): Unprotected vaginal or anal sex with a known HIV infected person or a casual partner, engaged in sex work for money or drugs, acquired a sexually transmitted disease, high risk partner currently or in the previous six months.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study (screening and Day -21) drug/alcohol screen.
* History of regular alcohol consumption within 6 months of the study as defined in the protocol.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Refrain from use of prescription or non-prescription drugs, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. If heparin is used during PK sampling, subjects with a history or sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* The subject has an underlying skin disease or disorder (i.e. infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria. Mild cases of localized acne or folliculitis are not exclusionary.)
* The subject has a tattoo or other dermatological condition overlying the gluteus and/or abdominal region which may interfere with interpretation of injection site reactions.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* History of clinically significant cardiovascular disease.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
GSK1265744 LAP safety and tolerability parameters including the collection of adverse events | approximately 25 weeks
GSK1265744 LAP safety and tolerability parameters including change from baseline in clinical laboratory safety assessments | approximately 25 weeks
  Hematology, Clinical Chemistry and Urinalysis
GSK1265744 LAP safety and tolerability parameters including change from baseline in electrocardiogram (ECG) measurements | approximately 25 weeks
GSK1265744 LAP safety and tolerability parameters including change from baseline in vital sign measurements | approximately 25 weeks
  Blood pressure and heart rate
TMC278 LA safety and tolerability parameters including the collection of adverse events | approximately 12 weeks
TMC278 LA safety and tolerability parameters including change from baseline in clinical laboratory safety assessments | approximately 12 weeks
  Hematology, Clinical Chemistry and Urinalysis
TMC278 LA safety and tolerability parameters including change from baseline in ECG measurements | approximately 12 weeks
TMC278 LA safety and tolerability parameters including change from baseline in vital sign measurements | approximately 12 weeks
  Blood pressure and heart rate
Composite of PK parameters following single and repeat dose intramuscular or subcutaneous administration | approximately 25 weeks
  Measurements include: area under the plasma concentration time curve over the dosing interval (AUC(0-t)), maximum observed concentration (Cmax), time to maximum observed concentration (tmax), concentration at the end of the dosing interval (Ct).
Composite of GSK1265744 pharmacokinetic parameters following repeat dose oral administration | approximately 25 weeks
  Measurements include: area under the plasma concentration time curve over the dosing interval (AUC(0-t)), maximum observed concentration (Cmax), time to maximum observed concentration (tmax), concentration at the end of the dosing interval (Ct).
Composite of TMC278 LA pharmacokinetic parameters following single and repeat dose intramuscular administration | approximately 12 weeks
  Measurements include: area under the plasma concentration time curve over the dosing interval (AUC(0-t)), maximum observed concentration (Cmax), time to maximum observed concentration (tmax), concentration at the end of the dosing interval (Ct).
GSK1265744 LAP safety and tolerability parameters including change from baseline for clinical chemistry assessments (ALT, AST, ALP, Total and Direct Bilirubin). | 52 weeks

SECONDARY OUTCOMES:
GSK1265744 oral formulation safety and tolerability parameters including the collection of adverse events | 21 days
GSK1265744 oral formulation safety and tolerability parameters including change from baseline in clinical laboratory safety assessments | 21 days
  Hematology, Clinical Chemistry and Urinalysis
GSK1265744 oral formulation safety and tolerability parameters including change from baseline in ECG measurements | 21 days
GSK1265744 oral formulation safety and tolerability parameters including change from baseline in vital sign measurements | 21 days
  Blood pressure and heart rate
Composite of PK parameters of GSK1265744 LAP and TMC278 LA | approximately 12 weeks
  Measurements include: apparent clearance (CL/FLAP) following single and repeat dose administration.
Composite of PK parameters following each dose administration at different dose levels for the assessment of dose proportionality and relative exposure | approximately 25 weeks
  Measurements include: GSK1265744 LAP AUC(0-t), Cmax, and Ct
Composite of PK parameters for GSK1265744 LAP | approximately 25 weeks
  Measurements include: apparent terminal phase half-life for LAP administration (t½), lambda z as a measure of absorption rate constant if data allow
Composite of PK parameters of TMC278 LA | approximately 12 weeks
  Measurements include: AUC(0-t), Cmax, and Ct in cohort 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (2):
- United States (2):
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Overland Park, Kansas